CLINICAL TRIAL: NCT01344746
Title: Leukotrienes Pathway in Chinese Children With Sleep-disordered Breathing
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Beijing Children's Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Shen Kunling/President, Beijing Children's Hospital
Other Study IDs: MISP 38608
Record Dates: First submitted 2011-04-28; First posted 2011-04-29 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2010-08

CONDITIONS: Sleep-disordered Breathing
Keywords: sleep-disordered breathing
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and adenotonsillar tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Snoring group: 1. Subjects with snoring and AHI ≥ 20 episodes/h (severe SDB).
  2. Snorers with AHI < 20 episodes/h and ≥ 5 episodes/h (moderate SDB)
  3. Snorers with AHI < 5 episodes/h and ≥ 1 episodes/h (mild SDB)
- Non-snoring group: * When testing serum and urinal samples, healthy children without snoring will be chosen as controls.
  * When testing lymphoid tissue samples, patients with recurrent infectious tonsillitis (at least five tonsillar infections in less than 6 months) but without snoring will be selected as controls before surgery and recruited to the study, because adenotonsillar tissue can't be obtained from normal children for obvious ethical reasons.

SUMMARY:
Our goals are to demonstrate an active leukotrienes (LTs) mediated inflammatory response is involved in pathophysiology of sleep-disordered breathing (SDB), and to provide a theoretical evidence for LTs modify therapy in treating pediatric patients with SDB.

The investigators have hypothesized that the pathophysiology of pediatric SDB involves specific systemic and local upper airway inflammatory response mediated by LTs.

1. LT concentration assays reveal higher levels in serum for both leukotriene B4 (LTB4) and cysteinyl leukotrienes (CysLTs) and in morning urine for LTE4 of SDB children, in comparison to healthy ones, and LTs productions emerge disease severity-dependent increases.

   There is a positive correlation between LTs production and other systemic markers such as neutrophil counts and high sensitive C-reactive protein (hsCRP).
2. Children with SDB have higher leukotriene receptor-1 (LT1-R) and leukotriene receptor-2 (LT2-R) expressions in adenotonsillar tissues of SDB children compared to recurrent infectious tonsillitis subjects.
3. Levels of LTs are positively correlated with body mass index (BMI) z-score, waist height ratio (WHtR), adenotonsillar size and polysomnography (PSG) indices including apnea-hypopnea index (AHI), obstructive apnea index (OAI), oxygen desaturation index (ODI), arousal index, percentage of time spend saturation lower than 90% (SLT90%) and negatively correlated with mean and minimal pulse oximetric saturation (SpO2), which indicates synergistic role of obesity and hypoxia are the determinants of LTs production in SDB.
4. In adenotonsillar mixed cell culture system, the addition of LTs can increase cellular proliferation rates and exhibit dose-dependent responses, whereas leukotriene receptor antagonists (LTRAs) elicit dose-dependent cellular reductions.

DETAILED DESCRIPTION:
Background:

SDB in children markedly differs from that seen in adults, in particular with respect to clinical manifestations, PSG (Polysomnography) findings, and treatment approaches. Pediatric SDB is due to a combination of increased upper airway resistance and repetitive pharyngeal collapsibility leading to intermittent hypoxemia and arousals during sleep. It is a common and highly prevalent disorder in pediatric age, affecting 4 to 11% of all children. If left untreated, it can result in serious morbid consequences including cardiovascular morbidity and neurocognitive dysfunction.

The etiology and pathophysiological mechanisms leading to SDB in childhood have not been clearly elucidated, but may include a complex interplay between anatomic (mainly adenotonsillar hypertrophy, ATH), neuromuscular factors and an underlying genetic predisposition toward the disease. However, more evidences have identified that both local airway and systemic inflammation also contribute to its pathogenesis.

Among major inflammatory mediators, leukotrienes (LTs) are a class of closely structurally related lipid compounds that derive from the 5-lipoxygenase pathway of arachidonic acid metabolism. The LTs family includes LTA4, LTB4 and LTC4/D4/E4 (cysLTs), all of which are potent leukocytes chemoattractants and activators. LTA4, an unstable intermediate, can be further metabolized to LTB4 or cysLTs. LTC4 and LTD4 both have very short half-lives, whereas LTE4 appears to be most stable. The effects of mediators occur after their interaction with receptors.

Recent investigations in western countries have revealed LTs may be involved in the pathogenesis of SDB, and accelerate the progress of the disease by exacerbating local inflammatory response, then promoting the proliferation of the upper airway lymphoid tissues. And in the later pediatric investigation, it was determined that LTs production emerged disease severity-dependent increases in exhaled breath condensate of SDB patients. Nevertheless, few studies have investigated the role of LTs in systemic inflammation of SDB, and whether LTs productions is a independent risk factor of SDB, or is a obesity-dependent or ATH -dependent risk factor of SDB remains controversial. Moreover, no research work in China has been carried out to investigate the LTs pathway in a large population of Chinese snoring children with SDB.

Participants:

Consecutive children referred to the sleep center for PSG due to symptoms of SDB from December 2009 to June 2010 were enrolled in the study. Normal age-, sex-, and weight-matched children without a history of snoring participated as control subjects, who were recruited from a community-based physical check-up activity.

Grouping:

Five groups of participants were formed:

1. Snoring group:

1. Subjects with snoring and AHI ≥ 20 episodes/h (severe SDB).
2. Snorers with AHI < 20 episodes/h and ≥ 5 episodes/h (moderate SDB)
3. Snorers with AHI < 5 episodes/h and ≥ 1 episodes/h (mild SDB)

2. Non-snoring control group:

* When testing serum and urinal samples, healthy children without snoring will be chosen as controls.
* When testing lymphoid tissue samples, patients with recurrent infectious tonsillitis (at least five tonsillar infections in less than 6 months) but without snoring will be selected as controls before surgery and recruited to the study, because adenotonsillar tissue can't be obtained from normal children for obvious ethical reasons.

The five study groups having at least 45 participants respectively will be compared regarding subjects' characteristics, PSG indices, metabolic and inflammatory variables.

Statistical Methods:

1. Data are presented as mean ± SD or median (interquartile range) depending on the distribution unless stated otherwise. PSG indexes, hsCRP values and LT concentrations will be log-transformed (natural logarithm) and SpO2 will be logit-transformed to correct for skewed distribution.
2. One-way analysis of variance followed by post hoc tests for pair comparisons (Bonferroni test) will be used for continuous variables and X2 test (Yates correction) for categorical characteristics. If data can't be transformed to approach normal distribution, Kruskal-Wallis test followed by nonparametric Bonferroni multiple comparison test will be applied.
3. Correlations will be analyzed without adjustment by using Pearson correlation or spearman rank test depending on data distribution. Partial correlation will be applied to assess the linear association of LTs concentrations with other systemic inflammatory marks and PSG indices after adjustment for covariates including age, glucose, lipids, and BMI z-score.
4. Stepwise multiple regressions will be performed to identify independent predictors of LTs production.
5. All statistical analyses will be conducted using statistical software (version 16.0; SPSS, Chicago, IL, USA). Using Dunnett's test, a two-tailed p value < 0.01 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were aged from 2 to 12 years ( 2 years ≤ subjects' age ≤ 12 years).
* Subjects who were in the presence of habitual snoring (snoring as reported by parents > 3 nights/week) and his/her history of habitual snoring were at least 3 months could be recruited in snoring group.
* Subjects who didn't have a history of snoring could be recruited as control subjects

Exclusion Criteria:

* Subjects who have cardiovascular, neuromuscular, craniofacial or genetic disorders; acute or chronic inflammation disease, e.g. asthma, allergic rhinitis or other allergies.
* Subjects who receive pharmacologic treatment including antibiotics, aspirin, nonsteroidal anti-inflammatory drugs, corticosteroids, and LTRAs within last 1 month.
* Subjects who already had undergone T&A in the past.
* Subjects who were receiving oral appliances or CPAP (Continuous Positive Airway Pressure ) treatment.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Consecutive children referred to the sleep center for PSG due to symptoms of SDB from December 2009 to June 2010 were enrolled in the study. Normal age-, sex-, and weight-matched children without a history of snoring participated as control subjects, who were recruited from a community-based physical check-up activity.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-11 (Estimated); Study Completion 2012-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kunling Shen, MD, Principal Investigator — Beijing Children's Hospital
Locations (1):
- Beijing Children's Hospital, Beijing, Beijing Municipality, China